CLINICAL TRIAL: NCT01019343
Title: Physiological Investigations of Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 100009; 10-N-0009
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-11-07

CONDITIONS: Parkinson's Disease; Tourette's Syndrome; Tic Disorders; Dystonia; Movement Disorders
Keywords: Magnetic Resonance Imaging (MRI); Magnetoencephalogram; Electroencephalogram (EEG); Transcranial Magnetic Stimulation (TMS); Motor Deficit
MeSH Terms: conditions — Parkinson Disease; Tourette Syndrome; Tic Disorders; Dystonia; Movement Disorders; Neurologic Manifestations | interventions — Transcranial Direct Current Stimulation; Exercise Test; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Placebo Comparator): Healthy Volunteers
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS); Device: Eye-tracking Device; Device: Pulsed vibrator; Other: Gait Trainer Treadmill (GTT); Other: Standard psychiatric scales SCID-I, YBOCS and SCI-OBS-lifetime and cognitive scales MMSE and MOCA; Device: iMobility; Device: QMAT; Diagnostic Test: Treadmill Test; Device: Arm Intellistretch Device; Procedure: Transcranial Sonography (TCS); Other: Behavioral tasks; Procedure: TMS single/paired pulse; Procedure: MEG; Procedure: EEG; Procedure: MRI techniques; Procedure: Peripheral Nerve Stimulation; Procedure: EMG; Procedure: Trancutaneous spinal direct current stimulation (tsDCS)
- Movement Disorder (Active Comparator): Subjects diagnosed with movement disorder
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS); Device: Eye-tracking Device; Device: Pulsed vibrator; Other: Gait Trainer Treadmill (GTT); Other: Standard psychiatric scales SCID-I, YBOCS and SCI-OBS-lifetime and cognitive scales MMSE and MOCA; Device: iMobility; Device: QMAT; Diagnostic Test: Treadmill Test; Device: Arm Intellistretch Device; Procedure: Transcranial Sonography (TCS); Other: Behavioral tasks; Procedure: TMS single/paired pulse; Procedure: MEG; Procedure: EEG; Procedure: MRI techniques; Procedure: Peripheral Nerve Stimulation; Procedure: EMG; Procedure: Trancutaneous spinal direct current stimulation (tsDCS)

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Transcranial direct current stimulation involves the application of weak direct currents, delivered between two surface electrodes, placed over the scalp.
Device: Eye-tracking Device — The purpose of this device is to assess eye movement. Participants may sit down in front of a computer screen or a real-world environment, stand on a treadmill, or lie down in an MRI scanner. Small infrared cameras attached to the cap or glasses will be positioned in front of their eyes. Eye tracking might be performed alone, or in conjunction with EEG, EMG, fMRI or treadmill. The eye- tracking device is FDA approved and commercially available.
Device: Pulsed vibrator — This device would be used in experiments to see if gait can be improved and, if so, what parameters of stimulation are optimal.
Other: Gait Trainer Treadmill (GTT) — The Gait Trainer is a specialized rehabilitation treadmill, which operates in both the forward and backwards mode allowing subjects to both train and undergo performance tasks in a relatively safe and expedient manner. The GTT is equipped with a mounted deck with built in sensors which monitors and records subjects gait speed, step length, right to left time distribution, and symmetry in real time in both forward and reverse modes.
Other: Standard psychiatric scales SCID-I, YBOCS and SCI-OBS-lifetime and cognitive scales MMSE and MOCA — Scales of motor function, cognitive function and psychiatric function are valuable supplements to clinical assessments of patients, giving quantitative information concerning these different aspects of brain function. Selected scales would be used only when potentially useful in a sub-study where such quantitative information would be correlated with a physiological or imaging result.
Device: iMobility — This test uses the iMobility system. iMobility Device is a small device designed to measure movement through sensors (test monitors) worn by a patient via Velcro straps around an ankle or wrist or worn as a pendant around the neck to lie over the sternum. The device is a nonsignificant risk device.The iMobility Device has been used before, in the same format with a similar paradigm, in previous NIH studies.
Device: QMAT — The purpose of this study is to assess the ability of the QMAT (quantitative motor assessment tool) to assess slowness of movement associated with Parkinson Disease. The QMAT device is FDA approved and has been used before, in the same format with a similar paradigm, in previous NIH studies.
Diagnostic Test: Treadmill Test — Subjects will be fitted in a weight support harness for safety. Sensors will be placed on the subject s shoes and harness. The sensors (VICON system) will be used to record their stride length, position and velocity as they walk on a treadmill. This system is a motion-tracking system that is designed to measure various aspects of a person s gait.
Device: Arm Intellistretch Device — The purpose of the Arm Intellistretch device is to objectively quantify wrist tone. It is used for rehabilitation applications in hospitals and office settings. Currently, rigidity is evaluated clinically using a subjective scale, zero to four and is part of the UPDRS. The Arm Intellistretch device is manufactured by Rehabtek, Inc., is FDA approved, and has been determined to be a non-significant risk device by the CNS IRB.
Procedure: Transcranial Sonography (TCS) — Transcranial sonography will be conducted by a physician in the Clinical Center using the Acuson Antares ultrasound machine. This techniques uses ultrasound signals to image the brain. It entails having the subject sit in a chair or lay in a bed while the sonographer places a lubricated 2-inch ultrasound probe over the skin of the temporal area just above the patient s ear. Ultrasound images are then recorded. The procedure is not invasive and will last about 45 minutes.
Other: Behavioral tasks — To assess the changes in cerebral physiology in the brain, subjects will be presented sensory stimuli (e.g., primary visual stimulation with flashing lights or checkerboard, auditory with tone or speech, or olfactory stimuli), or will be asked to perform non-exercise motor tasks (e.g., tapping of fingers, squeezing ball, moving joystick), to perform cognitive tasks such as a working memory task (e.g., n-back with or without catch rules, word finding), or to just rest or sleep.
Procedure: TMS single/paired pulse — For MEP acquisition during TMS, electrodes will be placed over the belly and the tendon of the distal muscles of the hand or foot and/or proximal muscles (see sub-section EMG 7.1.3.1 for the details of the procedure).
Procedure: MEG — MEG recordings will be performed together with experienced personnel in the NIMH MEG lab in the NMR center in Building 10. For these recording sessions, subjects will sit in a chair or lay down with a helmet placed over the head. The helmet used for MEG does not require the application of conductive gel. Scan times vary from 20 minutes to 2 hours.
Procedure: EEG — EEGs will be recorded by, or together with, experienced personnel in the HMCS EEG lab in Building 10, or in the NMR center.
Procedure: MRI techniques — MRI sub-studies will be conducted on 3.0 T or 7T units in the NMR Research Center. All volunteers will comply with the yearly requirement of a standard clinical diagnostic MRI scan of the head performed at 3.0T, to be submitted to the Diagnostic Radiology Department of the Clinical Center for interpretation. If the subject does not have a clinical scan performed within 12 month of the exam, a standard clinical MRI will be performed and reviewed before the research MR. The standard examination takes approximately 15 minutes to complete; after that, the research MR scans will be performed. Standard clinical MRI of the head will be repeated on an annual basis and read by the Diagnostic Radiology Department of the Clinical Center.
Procedure: Peripheral Nerve Stimulation — Constant-current, 0.1 to 0.5 ms square-wave single pulses of electrical stimulation will be delivered through standard bar electrodes to nerves of the upper limb or of the lower limb. To study somatosensory evoked potentials, for example, the stimulus intensity will be set at just above the motor threshold for evoking a slight limb movement. Location of the electrical stimulation will depend on the specific objective of the sub-study. Peripheral nerve stimulation might be delivered during other types of experiments as well.
Procedure: EMG — EMG measures the electrical activity of muscles. For our research purposes, only surface EMG will be used to measure the effects of central and peripheral nervous system stimulation. For surface EMG, electrodes will be coated with a conductive gel and taped to the skin. For motor evoked potential (MEP) acquisition during TMS, electrodes will be placed over the belly and the tendon of the distal muscles of the hand or foot and/or proximal muscles.
Procedure: Trancutaneous spinal direct current stimulation (tsDCS) — Direct current (DC) stimulation is a non invasive tool used to promote plasticity of the central nervous system. Recently, DC stimulation has been applied to the human spinal cord, and known as transcutaneous spinal direct current stimulation (tsDCS).

SUMMARY:
Background:

* Previous studies have given researchers information on how the brain controls movement, how people learn to make fine, skilled movements, and why some people have movement disorders. However, further research is needed to learn more about the causes of most movement disorders, such as Parkinson's disease.
* By using small, specialized studies to evaluate people with movement disorders and compare them with healthy volunteers, researchers hope to learn more about the changes in the brain and possible causes of movement disorders.

Objectives:

* To better understand how the brain controls movement.
* To learn more about movement disorders.
* To train movement disorder specialists.

Eligibility:

* Individuals 18 years of age or older who have had a movement disorder diagnosed by a neurologist and are able to participate based on the specific requirements of the small study.
* Healthy volunteers 18 years of age or older.

Design:

* Participants will have a screening visit with medical history, physical examination, and questionnaire to determine eligibility. Eligible participants will give consent to participate in up to seven additional outpatient visits for study procedures. The number of sessions and the procedures needed for participation depend on specific symptoms.
* Participants must avoid drinking alcohol or caffeinated drinks (sodas, coffee, and tea) for at least 2 days (48 hours) before each session.
* Potential studies may include magnetic resonance imaging (MRI) scans, functional MRI scans, electroencephalography, magnetoencephalography, transcranial magnetic stimulation, nerve and sensory stimulation, or movement and mental tasks during any of the above procedures.
* This study does not provide treatment for movement disorders. Participants will not have to stop any treatment in order to participate.

DETAILED DESCRIPTION:
Objectives

The purpose of this protocol is to improve understanding of the pathophysiology of movement disorders by performing small behavioral, electrophysiological and neuroimaging sub-studies. This will allow identifying dysfunction of the central nervous system that causes behavioral abnormalities seen in movement disorder patients. This will also help to determine potential diagnostic or therapeutic targets. Some sub-studies will require healthy volunteers. We will conduct:

* Pilot Sub-study (previously labeled as Small Pilot Sub-studies) Pilot sub-studies are exploratory in nature, in order to develop enough information to generate a hypothesis. The criterion for transition to a new full protocol will be a sufficient amount of information to generate a power analysis. There are no enrollment limitations for pilot sub-studies.Small substudies to pilot investigations for larger studies,
* Hypothesis-Testing Sub-study (previously labeled small number sSub-studies) is defined as a study with a specific hypothesis to be thattested that can be completed with a few subjects healthy volunteers or patients, , Hypothesis-testing sub-studies will undergo statistical and PIRC review after 6 subjects (if there is one group) or after 12 (six per arm) if two groups are studied before additional subjects are recruited. Together, the P.I. and PIRC will decide whether to continue the hypothesis sub-study with more subjects or if a new protocol is necessary. A memo requesting a review of hypothesis-testing sub-studies for possible additional enrollment will be sent to PIRC and the statistical reviewer. If the action to request accrual increase proceeds beyond PIRC to the IRB, then it needs to be submitted in the form of an amendment for prospective review/approval.
* Individual patient investigations that may increase knowledge of a disease process or be helpful in patient diagnosis,
* Training for investigators who do not have prior experience using electrophysiological and neuroimaging techniques,
* Technical development of new experimental paradigms.

This protocol includes only non-invasive techniques with minimal risk (MRI, EEG, MEG, peripheral nerve stimulation, TMS).

Study population

We intend to study 1200 healthy volunteers and 1000 patients with diagnoses of movement disorders.

Design

We will design small projects as ideas arise in our patient population that are pertinent to the theme of movement disorder pathophysiology. We will investigate patients with movement disorders or healthy volunteers in the resting state or while they perform simple motor or sensory tasks. If a small study leads to results of interest and if a larger population is necessary to reach statistical significance, a separate protocol will be submitted with a priori hypotheses, specific study design and power analysis adapted from the pilot or exploratory sub-studies performed in the present protocol.

Outcome measures

MRI: we will analyze measures such as the amplitude of the BOLD signal (fMRI); tractography between seed and target regions of interest (using DTI); morphometry of brain regions (using VBM); and different neurotransmitter levels in brain regions of interest (using MRS).

EEG and MEG: we will quantify measures such as event- or task-related potentials, synchronization/desynchronization, and coherence between sensors or sources located close to the brain areas of interest.

TMS: we will analyze measures such as MEP amplitude and central conduction time.

Behavioral measures: we will quantify measures such as reaction times to initiate movements, EMG patterns, movement kinematics (position, velocity, acceleration, curvature).

We may measure autonomic data during the course of the experiment (such as blood pressure, skin conductance, and respiratory rate) which would correlate to the outcome measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

INCLUSION CRITERIA FOR MOVEMENT DISORDER PATIENTS:

* Patients will either have a well-defined diagnosis or be a diagnostic dilemma, depending upon the sub-study
* Age 18 or older
* Able to give informed consent
* Agree to not drink caffeine or alcohol for 48 hours before certain study sessions because both agents can modify brain activity and may confound outcome measures.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Age 18 or older.
* Able to give informed consent.
* Agree to not drink caffeine or alcohol for 48 hours before certain study sessions because both agents may modify the activity of the brain during the study.

EXCLUSION CRITERIA:

EXCLUSION CRITERIA FOR MOVEMENT DISORDER PATIENTS:

* Have used illegal drugs within the past 6 months
* Have more than 7 alcoholic drinks a week in the case of a woman or 14 alcoholic drinks a week in the case of a man.
* Have had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures.
* Have a psychotic disorder, Bipolar Disorder or a current depressive episode.
* Have another neurologic disorder than a movement disorder
* Have had a head injury where there was a loss of consciousness for more than a few seconds.

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Have abnormal findings on a neurological examination that we will perform
* Have used illegal drugs within the past 6 months
* Have more than 7 alcoholic drinks a week in the case of a woman or 14 alcoholic drinks a week in the case of a man
* Have had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures.
* Have major depression or any major mental disorders (axis I disorders)
* Have had a head injury where there was a loss of consciousness for more than a few seconds.

ADDITIONAL EXCLUSION CRITERIA FOR MOVEMENT DISORDER PATIENTS AND HEALTHY VOLUNTEERS SPECIFICALLY FOR fMRI:

We will follow the NMR Center guidelines for MR safety.

Some of the exclusions are:

* Have non-MRI compatible metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or metal fragments in the eye as these make having an MRI unsafe.
* Unable to lie flat on the back for the expected length of the experiment up to 3 hours
* Have uncontrolled movements of the head
* Have an abnormality on the brain imaging or neurologic examination not related to the diagnosis
* Uncomfortable being in a small space for the expected length of the experiment up to 3 hours
* Pregnancy

ADDITIONAL EXCLUSION CRITERIA FOR MOVEMENT DISORDER PATIENTS AND HEALTHY VOLUNTEERS SPECIFICALLY FOR TMS:

* Have metal in the eye or skull area, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, metal fragments in the eye, as these make TMS unsafe. Having a cardiac pacemaker, intracardiac lines, implanted pumps or stimulators are also exclusion criteria.
* Have hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1273 (Actual)
Dates: Start 2009-12-08 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
MRI | throughout
  analyze measures such as the amplitude of the BOLD signal (fMRI); tractography between seed and target regions of interest (using DTI); morphometry of brain regions (using VBM); and different neurotransmitter levels in brain regions of interest (using MRS).
EEG and MEG | throughout
  quantify measures such as event- or task-related potentials, synchronization/desynchronization, and coherence between sensors or sources located close to the brain areas of interest.
TMS | throughout
  analyze measures such as MEP amplitude and central conduction time.
Behavioral measures | throughout
  quantify measures such as reaction times to initiate movements, EMG patterns, movement kinematics (position, velocity, acceleration, curvature), eye movement.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: Will be shared upon request after the IRB approves the sharing and after a data sharing agreement is in place.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-N-0009.html